CLINICAL TRIAL: NCT00164463
Title: TBTC Study 27/28 PK: Pharmacokinetic Issues in the Use of Moxifloxacin for Treatment of Tuberculosis
Brief Title: TBTC Study 27/28 PK: Moxifloxacin Pharmacokinetics During TB Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Bayer (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: William R. Mac Kenzie, MD / project officer, Tuberculosis Trial Consortium
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-4222
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin; Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin 400 mg po qd given 5 of 7 days per week
  Interventions: Drug: Moxifloxacin
- Isoniazid (Active Comparator): Isoniazid 300 mg po qd given 5/7 days per week
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Moxifloxacin — 400 mg po qd 5/7 days per week
  Arms: Moxifloxacin
Drug: Isoniazid — isoniazid 300 mg po qd 5/7 days per week
  Arms: Isoniazid

SUMMARY:
This substudy of TBTC Studies 27 and 28 compares 1) the pharmacokinetics of moxifloxacin alone versus moxifloxacin administered with rifampin in healthy volunteers and 2) the pharmacokinetics of moxifloxacin among patients with tuberculosis being treated with multidrug therapy (isoniazid or ethambutol, rifampin, and pyrazinamide) to those of healthy volunteers receiving moxifloxacin plus rifampin. It also evaluates the association between polymorphisms of MDR1 genotype (P-glycoprotein) and rifampin pharmacokinetic parameters, the effect of polymorphisms of MDR1 genotype and/or rifampin pharmacokinetics on isoniazid pharmacokinetic parameters adjusted for N-acetyltransferase genotype (NAT2), and determines by multivariate regression analyses the associations between moxifloxacin or rifampin pharmacokinetic parameters and markers of tuberculosis disease severity including the covariates of two-month culture positivity, cavitary lung disease, Body Mass Index, weight, duration of study treatment prior to PK, co-morbidities and C-reactive protein. Healthy volunteers and TB patients receive frequent scheduled blood draws during a 24 hour period after ingesting a dose of TB drugs.

ELIGIBILITY:
Inclusion Criteria:

For Healthy Volunteers:

* Provision of informed consent for the study.
* Age > 18 years.
* Willingness to be available for 2 weeks of DOT.
* Willingness to be admitted to a GCRC or hospital on two occasions.
* Women of child-bearing potential must agree to practice an adequate method of birth control. Barrier methods of contraception or abstinence from sexual activity are satisfactory methods.
* Willingness to have HIV testing done if documented results are not available. (A prior negative result must be obtained within one year and consists of a negative HIV ELISA. A positive result must be both a positive HIV ELISA and Western Blot, or a plasma HIV PCR RNA level greater than 5000 copies/ml).
* Laboratory screening (if not already available) within 30 days of the first PK admission:

  * Serum potassium within normal limits
  * Hematocrit > 35%
  * Absolute neutrophil count > 1000 /mm3
  * AST < 3 times the upper limit of normal
  * Bilirubin < 2 times the upper limit of normal
  * Creatinine < 2 times the upper limit of normal
* Eligible and enrolled for medical health care sponsored by the United States federal government (such as the Veterans Administration enrollment Priority 1 through 7, VHA Directive 2003-003).

For Patients with Tuberculosis Enrolled in TBTC Study 27 or Study 28:

* Any patient enrolled in TBTC Study 27 or Study 28 receiving a daily (5-7 days per week) regimen.
* Provision of informed consent for the study.
* Willingness to be admitted to a GCRC or hospital on one occasion.

Exclusion Criteria:

For Healthy Volunteers:

* Karnofsky score less than 90
* Pregnancy or breast-feeding. (A negative pregnancy test is required for women of childbearing potential within 14 days before the first dose of moxifloxacin.)
* Known allergy to any fluoroquinolone or rifamycin antibiotic
* Current or planned therapy during the study with drugs having unacceptable interactions with rifampin
* History of prolonged QT syndrome or current or planned therapy with quinidine, procainamide, amiodarone, sotalol, or ziprasidone during period of administration of moxifloxacin and for one week after treatment

For Patients with Tuberculosis Enrolled in TBTC Study 27 or Study 28:

* Severe anemia as defined by a hematocrit less than 25% (most recent value, measured within 30 days of the PK study).
* History of severe liver disease classified as Child Pugh Class C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Compare in healthy volunteers the pharmacokinetics of moxifloxacin alone versus moxifloxacin administered with rifampin. | study period
Compare the pharmacokinetics of moxifloxacin among patients with tuberculosis being treated with multidrug therapy (isoniazid or ethambutol, rifampin, and pyrazinamide) to those of healthy volunteers receiving moxifloxacin plus rifampin. | study period

SECONDARY OUTCOMES:
Determine variation of moxifloxacin pharmacokinetics (PK) among patients with pulmonary TB during treatment. | study period
Compare serum concentrations of isoniazid rifampin and pyrazinamide among patients being treated with moxifloxacin versus patients being treated with ethambutol as the fourth drug in multidrug treatment. | study period
Compare serum concentrations of rifampin, pyrazinamide and ethambutol among patients being treated with moxifloxacin versus patients being treated with isoniazid as the fourth drug | study period
Determine the association between polymorphisms of MDR1 genotype (P-glycoprotein) and rifampin PK parameters. | study period
Determine the effect of polymorphisms of MDR1 genotype and/or rifampin PK on isoniazid PK parameters adjusted for N-acetyltransferase genotype (NAT2). | study period
Determine the effects of polymorphisms of MDR1 and UGT genotypes on moxifloxacin PK parameters. | study period
Determine by multivariate regression analyses the associations between moxifloxacin or rifampin PK parameters and markers of disease severity. | study period

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Study Chair — VAMC and University of Texas Health Science Center San Antonio; William Burman, MD, Study Chair — Denver Public Health
Locations (8):
- United States (6):
  - University of Southern California Medical Center, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Veterans Administration Medical Center, Houston, Texas
  - Audie L Murphy Memorial Veterans Administration Medical Center, San Antonio, Texas
- University of British Columbia, Vancouver, British Columbia, Canada
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Result] Weiner M, Peloquin C, Burman W, Luo CC, Engle M, Prihoda TJ, Mac Kenzie WR, Bliven-Sizemore E, Johnson JL, Vernon A. Effects of tuberculosis, race, and human gene SLCO1B1 polymorphisms on rifampin concentrations. Antimicrob Agents Chemother. 2010 Oct;54(10):4192-200. doi: 10.1128/AAC.00353-10. Epub 2010 Jul 26. PMID 20660695
- [Result] Weiner M, Burman W, Luo CC, Peloquin CA, Engle M, Goldberg S, Agarwal V, Vernon A. Effects of rifampin and multidrug resistance gene polymorphism on concentrations of moxifloxacin. Antimicrob Agents Chemother. 2007 Aug;51(8):2861-6. doi: 10.1128/AAC.01621-06. Epub 2007 May 21. PMID 17517835
- [Derived] Weiner M, Gelfond J, Johnson-Pais TL, Engle M, Peloquin CA, Johnson JL, Sizemore EE, Mac Kenzie WR. Elevated Plasma Moxifloxacin Concentrations and SLCO1B1 g.-11187G>A Polymorphism in Adults with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2018 Apr 26;62(5):e01802-17. doi: 10.1128/AAC.01802-17. Print 2018 May. PMID 29463526